CLINICAL TRIAL: NCT02278510
Title: A Pilot Trial of Intraparenchymally-Administered Topotecan Using Convection-Enhanced Delivery (CED) in Patients With Suspected Recurrent/Progressive WHO Grade III or IV (High Grade) Glioma Requiring Stereotactic Biopsy
Brief Title: Topotecan Using Convection-Enhanced Delivery (CED) in High Grade Glioma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Michael Vogelbaum, MD, PhD (Other)
Collaborators: Infuseon Therapeutics, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Michael Vogelbaum, MD, PhD, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INFT1314; NCI-2014-02248 (Registry Identifier: CTRP)
Record Dates: First submitted 2014-10-28; First posted 2014-10-30 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Malignant Glioma; WHO Grade III or IV Recurrent Glioma
Keywords: topotecan; convection-enhanced delivery; CED; High Grade Glioma
MeSH Terms: conditions — Glioma; Lymphoma, Follicular | interventions — Topotecan; Gadolinium DTPA

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Direct infusion of topotecan (Experimental): The experimental Cleveland Multiport Catheter will be used to inject a chemotherapy, topotecan, and a contrast agent, gadolinium DTPA, into the high grade brain tumors of study participants
  Interventions: Drug: Topotecan; Drug: Gadolinium DTPA; Device: Cleveland Multiport Catheter

INTERVENTIONS:
Drug: Topotecan — Topotecan is a chemotherapy that is approved by the FDA to treat cancers. It is normally given by an intravenous injection, and not directly into a tumor. That is why it is considered to be an investigational drug for this study
Drug: Gadolinium DTPA — Gadolinium DTPA is a contrast agent which will be added to topotecan to allow the investigators to observe where topotecan goes in tumors. Gadolinium DTPA is approved by the FDA for intravenous injection during an MRI scan. It is not approved by the FDA for administration directly into a tumor.
Device: Cleveland Multiport Catheter — The Cleveland Multiport Catheter is a device that is not approved by the FDA and so it is classified as an investigational device. It has been designed to deliver drugs and other agents intended to treat cancers directly into the affected tissues. The Cleveland Multiport Catheter can be placed into a brain tumor only in the operating room. It is placed during an operation to perform a biopsy of brain tumors. Following the biopsy, a surgeon will place two catheters into the tumor with use of an image guided navigation system. Once each catheter has been placed, it will be secured into the scalp and the incision will be closed. The Cleveland Multiport Catheter will be left in place until the completion of the topotecan treatment.

SUMMARY:
Topotecan is a FDA-approved drug when given by intravenous injection, but it is not effective against brain tumors when given intravenously. The Cleveland Multiport Catheter is a new, investigational device that will be used to deliver topotecan directly into participants' brain tumors. One purpose of this study is to determine whether the Cleveland Multiport Catheter can be used effectively and safely to deliver topotecan directly into brain tumors. This study will also evaluate different doses of topotecan that can be delivered to a participant's brain tumor with use of the Cleveland Multiport Catheter, and it will also examine how their tumor responds to treatment with topotecan.

DETAILED DESCRIPTION:
This study will look at the way topotecan is injected into participant's tumor. A small amount of contrast dye (called gadolinium DTPA) will be added to topotecan before it is injected. Pictures will be taken of the tumor with an MRI machine. This will allow the investigators to see where in the tumor the topotecan has been injected. Issues related to patient selection, coordination with other therapeutic and palliative clinical options, and patient quality of life impact will be studied. Except for the infusion of topotecan and gadolinium DTPA into the tumor, and MRI imaging of the infusion process, all procedures and treatments participants will experience during the care of their brain tumor are non-investigational; the types of medical treatments, procedures, and tests they experience will be Standard of Care for patients with brain tumors.

Primary Objectives:

* To investigate by MR imaging the spatial and temporal distribution of topotecan in tumor and tumor-infiltrated brain administered by convection-enhanced delivery (CED) in patients with recurrent/progressive WHO grade III or IV (high grade) glioma (HGG) who have failed standard therapy comprising surgical biopsy and/or resection and adjuvant chemotherapy and radiotherapy
* To investigate by MR imaging the influence of the rate and topotecan concentration, on the spatial and temporal distribution of topotecan administered by CED in patients with recurrent/progressive HGG
* To evaluate the spatial and temporal distribution of topotecan, by MR imaging, when delivered into enhancing tumor tissue versus non-enhancing tumor tissue (as defined on pre-operative conventional MRI imaging with and without intravenous gadolinium)

Secondary Objectives:

* To investigate the extent to which backflow may be observed on MRI during CED-mediated delivery of topotecan
* To assess the safety, tolerability and toxicity profile of topotecan administered by CED using different doses and infusion rates
* To observe evidence of activity of single-agent topotecan administered by CED to patients with recurrent/progressive HGG who have failed standard therapy comprising surgical biopsy and/or resection and adjuvant chemotherapy and radiotherapy

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of supratentorial WHO Grade III or IV (High Grade Glioma) that has undergone surgical biopsy or resection followed by adjuvant chemoradiotherapy, that has evidence of recurrence or progression based on imaging studies and a stereotactic biopsy is indicated for confirmation of recurrence/progression
* Karnofsky Performance Status 70-100
* MRI demonstration of a stereotactically accessible enhancing mass of less than 40cm3 that does not require resection to relieve clinically significant mass effect
* Patient understands the procedures and agrees to comply with the study requirements by providing written informed consent

Laboratory values within the following ranges:

* Absolute neutrophil count (ANC)≥1,500/microliter
* Platelet count≥100,000/microliter
* Hemoglobin≥10g/dL
* Normal PT/PTT
* Estimated glomerular filtration rate (eGFR) of at least 50mL/min

Exclusion Criteria:

* Patient is mentally or legally incapacitated at the time of the study
* Known HIV(+) or has been diagnosed with AIDS
* Participation in another investigational drug study in the prior 4 weeks
* Positive pregnancy test in a female
* Patient, in the opinion of the investigator, is likely to be poorly compliant
* Diffuse subependymal or CSF disease
* Tumors involving the cerebellum
* Tumor enhancement involving both hemispheres
* Active infection requiring treatment
* Unexplained febrile illness
* Radiation or chemotherapy within 4 weeks of enrollment
* Systemic diseases associated with unacceptable anesthesia or operative risk
* Inability to undergo magnetic resonance imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-12-09 (Actual); Primary Completion 2015-11-10 (Actual); Study Completion 2015-11-10 (Actual)

PRIMARY OUTCOMES:
Spatial distribution of topotecan | 24 weeks
  Determination of the spatial distribution of intraparenchymally-administered topotecan over time using a gadolinium-based contrast agent, volumetric magnetic resonance imaging, and three-dimensional image reconstruction
Number of catheter- and/or drug-related complications | 24 weeks
  The overall number of catheter- and/or drug-related complications occurring intra-operatively, post-operatively, or following catheter removal

SECONDARY OUTCOMES:
Objective response rate of subjects given topotecan | 24 weeks
  The mean objective response rate to using the Response Assessment in Neuro-Oncology (RANO) criteria for single-agent topotecan in recurrent/progressive HGG administered via CED.
Median progression-free survival of HGG subjects given topotecan | 24 weeks
  The median progression-free survival of subjects in months using the Response Assessment in Neuro-Oncology (RANO) criteria for single-agent topotecan in recurrent/progressive GBM administered via CED.
Median overall survival of HGG subjects given topotecan | 24 weeks
  The median overall survival of subjects in months using the Response Assessment in Neuro-Oncology (RANO) criteria for single-agent topotecan in recurrent/progressive GBM administered via CED.
Proportion of progression free HGG subjects given topotecan | 24 weeks
  The proportion of subjects without disease progression using the Response Assessment in Neuro-Oncology (RANO) criteria for single-agent topotecan in recurrent/progressive GBM administered via CED.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Vogelbaum, MD, PhD, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Vogelbaum MA, Brewer C, Barnett GH, Mohammadi AM, Peereboom DM, Ahluwalia MS, Gao S. First-in-human evaluation of the Cleveland Multiport Catheter for convection-enhanced delivery of topotecan in recurrent high-grade glioma: results of pilot trial 1. J Neurosurg. 2018 Apr 13;130(2):476-485. doi: 10.3171/2017.10.JNS171845. Print 2019 Feb 1. PMID 29652233